CLINICAL TRIAL: NCT03552367
Title: Efficacy of a Structured Exercise Prescription Program Over Anthropometric, Metabolic and Fitness Parameters in Obese Children and Adolescents Included in a Multicomponent Lifestyle Intervention Program. Randomized Clinical Trial
Brief Title: Structured Exercise Prescription Program in Obese Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other); Fundacion Sertull (Unknown); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Nayely Garibay Nieto, Head of the Child and Adolescent Obesity Clinic, Hospital General de México Dr. Eduardo Liceaga
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DI/17/311/03/028
Record Dates: First submitted 2018-04-24; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Exercise; Cardiovascular Risk Factor; Liver Diseases; Metabolic Syndrome; Childhood Obesity
Keywords: Obesity; Children; Non-alcoholic fatty acid liver disease; Exercise; Metabolic syndrome; Cardiovascular risk
MeSH Terms: conditions — Obesity; Motor Activity; Liver Diseases; Metabolic Syndrome; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Randomized open clinical trial
Masking Description: This is an open-label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized structured exercise (Experimental): This group will be enrolled in a multicomponent program for obese children (8-12 years old) that includes intervention workshops concerning nutrition, emotional factors, cognitive therapy and personalized structured exercise prescription that will be offered on-site and online and monitored through the use of heart rate monitoring devices. The type of exercise offered to patients in this arm is precisely designed for obese patients according to age and physical fitness parameters.
  Intervention: Non-personalized non-structured exercise
  Interventions: Other: Personalized structured exercise program
- Non-personalized non-structured exercise (Active Comparator): This group will be enrolled in a multicomponent program for obese children (8-12 years old) that includes intervention workshops concerning nutrition, emotional factors, cognitive therapy and non-personalized non-structured exercise prescription Intervention: Non-personalized non-structured exercise
  Interventions: Other: Non personalized non-structured exercise program

INTERVENTIONS:
Other: Personalized structured exercise program — The type of exercise offered to patients in this arm is precisely designed for obese patients according to age and physical fitness parameters. Patients are monitored using a heart rate monitor to evaluate treatment adherence and compliance
  Other Names: Structured exercise
  Arms: Personalized structured exercise
Other: Non personalized non-structured exercise program — The type of exercise is non-structured and patients' heart rate is not monitored. Patients receive exercise recommendations without any personalization according to their fitness parameters
  Other Names: Non-structured exercise
  Arms: Non-personalized non-structured exercise

SUMMARY:
This controlled clinical trial aims to compare the effects of a multicomponent program that includes structured personalized exercise prescription in children with obesity with a control group that will be enrolled in a multicomponent program without structured personalized exercise prescription. All children will be followed for a period of 6 months.

The parameters that will be evaluated between groups are physical fitness, anthropometry, metabolic (glucose oral tolerance curve, lipids, HOMA-IR, ISI-MATSUDA), early cardiovascular damage, inflammatory biomarkers, anxiety and depression scores, and allelic variants related to physical fitness.

DETAILED DESCRIPTION:
This controlled clinical trial aims to compare the effects of a multicomponent program that includes structured personalized exercise prescription in children with obesity (study group) with a control group that will be enrolled in a multicomponent program without structured personalized exercise prescription. All children will be followed for a period of 6 months.

The parameters that will be evaluated between groups are physical fitness (measured by VO2max, ECG at rest, biomechanics and dynamometry), anthropometric measurements (weight height, BMI, plicometry, bioimpedance, metabolic (glucose oral tolerance curve, lipids, HOMA-IR, ISI-MATSUDA), early cardiovascular damage (carotid intima-media thickness, atherogenic dyslipidemia), inflammatory biomarkers (leptin, adiponectin, IL-17, IL-10, INF-gamma, IL-6, IL-12, y TNF-alpha), anxiety and depression scores evaluated with Child Depression Inventory (CID) and -Trait Anxiety Inventory for Children (STAI-CH), and allelic variants related to physical fitness (ACTN, TRH2 y FTO).

ELIGIBILITY:
Inclusion Criteria: Patients with BMI ≥ Pc 95 and < 35kg/m2 Both sexes Accepts to participate and signs informed consent

Exclusion Criteria:

Presence of endocrine disease including type I and II diabetes mellitus Presence of arterial hypertension Presence of primary dyslipidemia Presence of infections at moment of enrollment Presence of systemic disease Presence of genetic disorder Medical treatment that may interfere with lipid or glucose metabolism Prolonged or acute immobilization Participated in a previous similar intervention

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
VO2 max | 6 months
  Changes in VO2 max as fitness indicator
OGTT | 6 months
  Oral glucose tolerance test

SECONDARY OUTCOMES:
BMI | 6 months
  BMI zScore
AST | 6 months
  AST
ALT | 6 months
  ALT
GGT | 6 months
  GGT
Leptin | 6 months
  Leptin
Adiponectin | 6 months
  Adiponectin
Lean body mass | 6 months
  Lean body mass

CONTACTS AND LOCATIONS:
Overall Officials: Nayely Garibay Nieto, MD MSc, Principal Investigator — Director Child and Adolescent Obesity Clinic
Locations (1):
- Hospital General de Mexico Eduardo Liceaga, Mexico City, Del. Cuauhtemoc, Mexico

IPD SHARING:
Plan to Share IPD: No
Not until first article is published

REFERENCES:
- [Background] Krebs NF, Himes JH, Jacobson D, Nicklas TA, Guilday P, Styne D. Assessment of child and adolescent overweight and obesity. Pediatrics. 2007 Dec;120 Suppl 4:S193-228. doi: 10.1542/peds.2007-2329D. PMID 18055652
- [Background] American Dietetic Association (ADA). Position of the American Dietetic Association: individual-, family-, school-, and community-based interventions for pediatric overweight. J Am Diet Assoc. 2006 Jun;106(6):925-45. doi: 10.1016/j.jada.2006.03.001. PMID 16812927
- [Background] Kelley GA, Kelley KS. Exercise and BMI z-score in overweight and obese children and adolescents: protocol for a systematic review and network meta-analysis of randomised trials. BMJ Open. 2016 Apr 15;6(4):e011258. doi: 10.1136/bmjopen-2016-011258. PMID 27084289
- [Background] Kelley GA, Kelley KS, Pate RR. Exercise and BMI z-score in Overweight and Obese Children and Adolescents: A Systematic Review and Network Meta-Analysis of Randomized Trials. J Evid Based Med. 2017 May;10(2):108-128. doi: 10.1111/jebm.12228. PMID 27792271
- [Background] Lison JF, Real-Montes JM, Torro I, Arguisuelas MD, Alvarez-Pitti J, Martinez-Gramage J, Aguilar F, Lurbe E. Exercise intervention in childhood obesity: a randomized controlled trial comparing hospital-versus home-based groups. Acad Pediatr. 2012 Jul-Aug;12(4):319-25. doi: 10.1016/j.acap.2012.03.003. Epub 2012 May 26. PMID 22634075